CLINICAL TRIAL: NCT06095687
Title: Investigating the Effectiveness of Mindfulness Meditation and Clinical Hypnosis for Injury-related Pain Management in Elite Athletes
Brief Title: Mind-body Therapies for Injury-related Pain Management in Elite Athletes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of access to intended participant pool due to investigator changes
Sponsor: The University of Queensland (Other)
Collaborators: University of Alabama, Tuscaloosa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UniQueensland
Record Dates: First submitted 2023-10-11; First posted 2023-10-23 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2023-10

CONDITIONS: Pain, Acute
Keywords: Mindfulness meditation; Clinical hypnosis; Elite athletes
MeSH Terms: conditions — Acute Pain | interventions — Mindfulness; Hypnosis

STUDY DESIGN:
Intervention Model Description: Replicated single case experimental design
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blind to participant condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Meditation (Active Comparator): Condition 1, Mindfulness Meditation (MM): The MM recording will be adapted from Day (2017). It will first instruct the listener to anchor attention on the breath while being mindfully aware of any physical sensations that arise throughout the body. The listener is then encouraged to explore sensations with non-judgmental attentiveness, without attempts to change the sensation in any way. This will implicitly provide training in mindful acceptance. Finally, the listener is instructed to simply label any thinking that arises as "thinking", before returning to the object of the meditation.
  Interventions: Behavioral: Mindfulness Meditation
- Clinical Hypnosis (Active Comparator): Condition 2, Clinical Hypnosis (HYP): The HYP recording will be adapted from Jensen (2011). It will take the listener through a standardised self-hypnosis practice that includes an induction, followed by tailored suggestions. Specifically, the HYP session aims to take the listener through four basic ideas: 1) an induction to get the individual into a state of readiness to accept new ideas; 2) instructions to go to a favourite place to deepen the induction and provide a context for feeling heat while being relaxed; 3) linking suggestions for reducing automatic behavioural inhibition system and behavioural activation system (BIS-BAS) activation in response to stressors and enhancing awareness of when to activate each system; 4) suggestions that target enhancing self-confidence in pain management, well-being and the rehabilitation process; and 5) alerting.
  Interventions: Behavioral: Clinical Hypnosis

INTERVENTIONS:
Behavioral: Mindfulness Meditation — Five, 20-minute audio-recorded training sessions of mindfulness of breath and body meditation, practiced over consecutive days, delivered remotely via Qualtrics.
  Arms: Mindfulness Meditation
Behavioral: Clinical Hypnosis — Five, 20-minute audio-recorded training sessions of clinical hypnosis with suggestions targeting pain management, practiced over consecutive days, delivered remotely via Qualtrics.
  Arms: Clinical Hypnosis

SUMMARY:
This study will utilize a replicated single case experimental design (RSCD) to investigate the effectiveness of a brief mindfulness meditation (MM) vs clinical hypnosis (HYP) training for improving pain in injured elite athletes. The primary outcome is change in pain intensity. It is hypothesized that: (1) both treatments will engender clinically meaningful improvement in pain intensity; (2) change in cognitive processes will be a unique mechanism underlying improved pain outcome in MM, and (3) change in cognitive content will be a unique mechanism underlying improved pain outcome in HYP. This research program has the potential to reduce athletes' uncertainty around pain, time out with injury and improve pain management during rehabilitation and recovery from injury.

DETAILED DESCRIPTION:
The proposed program of research will utilize our current understanding of the Behavioral Inhibition System and Behavioral Activation System (BIS-BAS) model of pain and mind-body therapies and apply it to pain experienced by injured elite athletes. This study will be a replicated single case experimental design (RSCD), which will investigate the effectiveness of a brief mindfulness meditation (MM) vs clinical hypnosis (HYP) training for improving the primary outcome of pain intensity in injured elite athletes. It will also investigate the potential mechanism role of change in cognitive content and cognitive processes in underlying the effects of these mind-body therapies. It is hypothesized that: (1) both treatments will engender clinically meaningful improvement in pain intensity; (2) change in cognitive processes will be a unique mechanism underlying improved pain outcome in MM, and (3) change in cognitive content will be a unique mechanism underlying improved pain outcome in HYP. This research program has the potential to reduce athletes' uncertainty around pain, time out with injury and improve pain management during rehabilitation and recovery from injury.

ELIGIBILITY:
Inclusion Criteria:

* be an elite athlete (i.e., competing at international or division 1 varsity level),
* currently have a sport or exercise-related injury that resulted in an average pain intensity greater than or equal to 3 on a 0-10 numerical rating scale in the past week, and for which the predicted recovery time at the point of study enrolment is greater than 5 weeks,
* Be 18 or over.
* Read, speak, and understand the English language.
* Have access to the internet on a computer or smartphone.
* Have access to a set of headphones.
* Be willing to be randomly assigned to both conditions and listen to five 20-minute treatment sessions.
* Be willing to participate in a daily survey for 25 consecutive days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-05-05 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) of Current Pain Intensity | Assessed online daily during randomized baseline length of 5, 10 or 15 days, 5 day treatment period, and randomized post-treatment phase of 5, 10 or 15 days of assessment
  Change in pain intensity will be measured using a 0-10 numerical rating scale (NRS) of average pain in the past 24 hours. Participants will be asked to choose a number from 0-10 that best represents their pain intensity. Higher scores indicate higher levels of self-reported pain intensity.

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) of Current Pain Unpleasantness | Assessed online daily during randomized baseline length of 5, 10 or 15 days, 5 day treatment period, and randomized post-treatment phase of 5, 10 or 15 days of assessment
  Change in pain unpleasantness will be measured using a 0-10 numerical rating scale (NRS) of average pain unpleasantness in the past 24 hours. Participants will be asked to choose a number from 0-10 that best represents their pain unpleasantness. Higher scores indicate higher levels of self-reported pain unpleasantness.

OTHER OUTCOMES:
Depression Anxiety Stress Scale, 9-item SF, Stress Subscale | Assessed online daily during randomized baseline length of 5, 10 or 15 days, 5 day treatment period, and randomized post-treatment phase of 5, 10 or 15 days of assessment
  Change in general stress will be measured, with participants indicating how often they experience certain stress responses on a scale from 0 (never) to 3 (almost always).
Positive and Negative Affect Schedule - Serene Affect Subscale | Assessed online daily during randomized baseline length of 5, 10 or 15 days, 5 day treatment period, and randomized post-treatment phase of 5, 10 or 15 days of assessment
  Change in serene affect will be measured with participants rating three adjectives describing serenity affect (i.e., relaxed, at ease, calm) on a 5-point scale ranging from 1 (very slightly or not at all) to 5 (extremely).

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Queensland, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No
Aggregate data will be made available for research purposes upon reasonable request once the data are published (within a time period of 5-years), with a data sharing agreement put in place.